CLINICAL TRIAL: NCT02155738
Title: The Impact of IV Acetaminophen on Postoperative Pain in Women Undergoing Pelvic Organ Prolapse Repair: A Double-Blind Randomized Placebo Controlled Trial
Brief Title: IV Acetaminophen for Postoperative Pain After Pelvic Organ Prolapse Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Halina M Zyczynski, MD (Other)
Responsible Party: Sponsor-Investigator, Halina M Zyczynski, MD, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PFD-C-14-009
Record Dates: First submitted 2014-05-29; First posted 2014-06-04 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-10

CONDITIONS: Pelvic Organ Prolapse
Keywords: IV acetaminophen; Postoperative pain; Pelvic organ prolapse surgery; Pelvic organ prolapse repair
MeSH Terms: conditions — Pelvic Organ Prolapse; Pain, Postoperative | interventions — Acetaminophen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 100 cc of normal saline administered intravenously 10-30 minutes prior to anesthesia induction on the day of surgery.
  Interventions: Drug: IV normal saline
- IV Acetaminophen (Experimental): 100 cc of Acetaminophen (1000mg/100mL) administered intravenously 10-30 minutes prior to anesthesia induction on the day of surgery.
  Interventions: Drug: IV Acetaminophen

INTERVENTIONS:
Drug: IV Acetaminophen
  Other Names: Ofirmev
  Arms: IV Acetaminophen
Drug: IV normal saline — IV normal saline
  Other Names: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether preoperative IV Acetaminophen reduces postoperative pain and narcotic consumption in women undergoing surgical repair of pelvic organ prolapse.

DETAILED DESCRIPTION:
This randomized controlled trial of IV Acetaminophen compared to placebo will evaluate the effect of preoperative IV Acetaminophen on postoperative pain scores and narcotic requirements in women undergoing surgical repair of pelvic organ prolapse. 204 women will randomly receive 1000 mg of IV Acetaminophen or saline preoperatively within 30 minutes of surgical incision. Subjects will be offered narcotic and non-narcotic pain medications as needed during the postoperative period. Visual analogue pain scales (VAS) will be obtained at 4, 8, 12, 16, 20 and 24 hours postoperatively. Narcotic consumption will be recorded in morphine-equivalents. We hypothesize that women receiving IV Acetaminophen will have lower VAS scores and decreased narcotic requirements compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years of age
* scheduled to undergo surgery for POP via a vaginal or minimally invasive (laparoscopic/robotic) route at the University of Pittsburgh Medical Center
* women anticipated to have a hospital stay ≥24 hours

Exclusion Criteria:

* allergy/intolerance to acetaminophen
* hepatic dysfunction
* significant alcohol use - defined as patient reported consumption of more than 7 standard drinks per week and/or 3 drinks per day

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2014-07; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Magee-Womens Hospital of the University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Turner LC, Zyczynski HM, Shepherd JP. Intravenous Acetaminophen Before Pelvic Organ Prolapse Repair: A Randomized Controlled Trial. Obstet Gynecol. 2019 Mar;133(3):492-502. doi: 10.1097/AOG.0000000000003102. PMID 30741813

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were recruited form the Urogynecology offices of the University of Pittsburgh Medical Center (UPMC) and Allegheny Health Network (AHN) from July 2014 - August 2017.
Groups:
- Vaginal Surgery - Placebo: 100 cc of normal saline administered intravenously 10-30 minutes prior to anesthesia induction on the day of surgery.
  IV normal saline
  These subjects underwent vaginal surgery.
- Vaginal Surgery - IV Acetaminophen: 100 cc of Acetaminophen (1000mg/100mL) administered intravenously 10-30 minutes prior to anesthesia induction on the day of surgery.
  IV Acetaminophen
  These subjects underwent vaginal surgery.
- Laparoscopic Surgery - Placebo: 100 cc of normal saline administered intravenously 10-30 minutes prior to anesthesia induction on the day of surgery.
  IV normal saline
  These subjects underwent laparoscopic surgery.
- Laparoscopic Surgery - IV Acetaminophen: 100 cc of Acetaminophen (1000mg/100mL) administered intravenously 10-30 minutes prior to anesthesia induction on the day of surgery.
  IV Acetaminophen
  These subjects underwent laparoscopic surgery.
Period: Overall Study
Arm/Group | Vaginal Surgery - Placebo | Vaginal Surgery - IV Acetaminophen | Laparoscopic Surgery - Placebo | Laparoscopic Surgery - IV Acetaminophen
Started | 50 | 52 | 51 | 51
Completed | 49 | 52 | 51 | 50
Not Completed | 1 | 0 | 0 | 1
Not completed — Missing critical information | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: One subject in the Vaginal Surgery - Placebo group, and one subject in the Laparoscopic Surgery - IV Acetaminophen group did not complete the study. (Missing critical information: (1) information from the pharmacy regarding group assignment; (2) signed informed consent form.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaginal Surgery - Placebo | Vaginal Surgery - IV Acetaminophen | Laparoscopic Surgery - Placebo | Laparoscopic Surgery - IV Acetaminophen | Total
Number analyzed (Participants) | 49 | 52 | 51 | 50 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.24 (10.87) | 70.5 (9.20) | 60.22 (8.00) | 62.08 (7.00) | 65.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 52 | 51 | 50 | 202
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 1 | 2 | 0 | 1 | 4
  Caucasian | 47 | 50 | 51 | 48 | 196
  Other | 0 | 0 | 0 | 1 | 1
  Missing | 1 | 0 | 0 | 0 | 1
Postmenopausal [Count of Participants; unit: Participants] | 43 | 49 | 44 | 45 | 181
Current Smoker [Count of Participants; unit: Participants] | 3 | 2 | 2 | 1 | 8
Parity [Median (Inter-Quartile Range); unit: births] — Parity refers to the number of times the subject gave birth to a baby more than 20 weeks gestation. Parity is expressed as a whole number.
  births | 2 [2 to 3] | 2 [2 to 3] | 2 [2 to 3] | 2 [2 to 3] | 2 [2 to 3]
Baseline POPQ Stage [Count of Participants; unit: Participants] — POP-Q Stage is the Pelvic Organ Prolapse Quantification Stage. This is a whole number which refers to the extend of the prolapse, and how far past the hymen it extends. POP-Q Stage is a whole number between 1 and 4. Stage 1 is prolapse which is fully contained within the vagina and above the hymen. Stage 4 is prolapse which extends at least 3 cm beyond the hymen.
  Participants
    Stage II | 8 | 7 | 8 | 5 | 28
    Stage III | 35 | 37 | 42 | 37 | 151
    Stage IV | 5 | 7 | 1 | 8 | 21
    Missing | 1 | 1 | 0 | 0 | 2
Baseline VAS Pain Score [Mean (Standard Deviation); unit: units on a scale] — VAS or Visual Analog Score is a quantitative measure, in this study, of pain that the subject is currently experiencing. The VAS is presented as a straight line which measures 100mm. The subject is instructed to mark an 'X' through this line reflecting the amount of pain that they are currently experiencing. Zero would indicate no pain, while '100' would indicate the most severe pain ever. Thus the total range for this scale would be 0-100 mm. Higher values indicate more pain; lower value indicate less pain.
  units on a scale | 7.32 (15.73) | 3.41 (8.71) | 5.57 (15.60) | 6.91 (12.75) | 5.75 (13.45)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Postoperative Pain
Description: VAS or Visual Analog Score is a quantitative measure, in this study, of pain that the subject is currently experiencing. The VAS is presented as a straight line which measures 100mm. The subject is instructed to mark an 'X' through this line reflecting the amount of pain that they are currently experiencing. Zero would indicate no pain, while '100' would indicate the most severe pain ever. Thus the total range for this scale would be 0-100 mm. Higher values indicate more pain; lower value indicate less pain.
  For this outcome measure, the VAS scores from Baseline and the VAS scores from 24 hours after the end of surgery are being used. The change from baseline in postoperative pain equals the 24 hour VAS score minus the baseline VAS score.
  The Change from Baseline would be the 24-hour VAS score minus the Baseline VAS score. Higher values indicate more pain; lower values indicate less pain.
Time Frame: 24 hours
Population: The number of participants analyzed is less than the total starting the study in each group; data is missing. Missing data indicates that a 24 hour VAS was not obtained from the subject.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vaginal Surgery - Placebo | Vaginal Surgery - IV Acetaminophen | Laparoscopic Surgery - Placebo | Laparoscopic Surgery - IV Acetaminophen
Number analyzed (Participants) | 44 | 41 | 41 | 36
units on a scale | 20.5 (23.1) | 29.2 (28.3) | 20.7 (24.6) | 20.1 (25.7)
Statistical Analysis 1: Comparison: Vaginal Surgery - Placebo vs Vaginal Surgery - IV Acetaminophen vs Laparoscopic Surgery - Placebo vs Laparoscopic Surgery - IV Acetaminophen; Aim 1: Quantify the impact of IV acetaminophen on 1a) postoperative pain scores ... 1a) To achieve this aim, we will measure the degree of postoperative pain using visual analog scales (VAS) at multiple specified time points throughout the postoperative period; we report on change from Baseline VAS at 24 Hours Postop. Null Hypothesis is that there is no difference between subgroups in VAS scores. Sample size was determined considering significant differences in VAS scores; Test type: Superiority; p < 0.05, Mixed Models Analysis

2. Primary Outcome: Cumulative Narcotic Consumption Over the First 24 Hours
Description: Equianalgesic dosage tables will be used to convert intra- and postoperative narcotics into morphine equivalents to compare narcotic requirements for the first week after surgery. Higher numbers indicate higher narcotic usage.
Time Frame: First 24 hours
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Vaginal Surgery - Placebo | Vaginal Surgery - IV Acetaminophen | Laparoscopic Surgery - Placebo | Laparoscopic Surgery - IV Acetaminophen
Number analyzed (Participants) | 49 | 52 | 51 | 50
mg | 32.5 (24.7) | 31.6 (23.6) | 47.4 (24.2) | 44.5 (24.2)
Statistical Analysis 1: Comparison: Vaginal Surgery - Placebo vs Vaginal Surgery - IV Acetaminophen vs Laparoscopic Surgery - Placebo vs Laparoscopic Surgery - IV Acetaminophen; 1b) We will use equianalgesic dosage tables to convert intra- and postoperative narcotics into morphine equivalents to compare narcotic requirements for the first week after surgery. We hypothesize that those patients receiving preemptive IV acetaminophen will have lower postoperative VAS scores and reduced narcotic requirements compared to placebo; Test type: Superiority; p < 0.05, t-test, 2 sided

3. Secondary Outcome: Interference of Pain With Physical, Mental and Social Activities
Description: Interference of pain with physical, mental and social activities will be measured by the Patient Reported Outcomes Measures Information Systems-Pain Interference-Short Form 8a (PROMIS PI-SF-8a) administered on POD#7.
  This instrument measures the self reported consequences of pain on relevant aspects of one's life. This scale is considered to be universal rather than disease specific. Each question has five response options ranging in value from 1-5. The total raw score for the scale is the sum of all values. The total raw score can range from 8-40. All questions much be answered to obtain a valid score.
  A higher PROMIS score indicates more 'hurt' or pain.
Time Frame: 1 week
Population: The number of participants analyzed is less than the total starting the study in each group; data is missing. Missing data indicates that the PROMIS PI-SF-8A was not received from the subject.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vaginal Surgery - Placebo | Vaginal Surgery - IV Acetaminophen | Laparoscopic Surgery - Placebo | Laparoscopic Surgery - IV Acetaminophen
Number analyzed (Participants) | 41 | 33 | 44 | 40
units on a scale | 18.4 (0.15) | 22.0 (11.9) | 22.9 (8.1) | 25.2 (9.4)

ADVERSE EVENTS:
Time Frame: AEs were collected from day of surgery until 6 weeks postop.
Description: SAEs were defined a priori as readmissions to the hospital for any reason within 6 weeks of surgery. All subject medical records were reviewed to discover these events.
Arm/Group | Vaginal Surgery - Placebo | Vaginal Surgery - IV Acetaminophen | Laparoscopic Surgery - Placebo | Laparoscopic Surgery - IV Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/52 | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 1/49 | 1/52 | 0/51 | 3/50
Other Adverse Events (participants affected / at risk) | 0/49 | 0/52 | 0/51 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaginal Surgery - Placebo (N=49) | Vaginal Surgery - IV Acetaminophen (N=52) | Laparoscopic Surgery - Placebo (N=51) | Laparoscopic Surgery - IV Acetaminophen (N=50)
Readmission within 6 weeks of surgery (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 3 (3) — Any readmission within 6 weeks of surgery. Medical records for all subjects were reviewed to discover these events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT02155738/Prot_SAP_000.pdf